CLINICAL TRIAL: NCT04685057
Title: Probiotics as a Long-term Treatment Strategy for Prader-Willi Syndrome
Brief Title: Probiotic Treatment for Prader-Willi Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PIC-194-20
Record Dates: First submitted 2020-12-02; First posted 2020-12-28 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-01

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): This arm will receive placebo for 6 months then probiotic for 6 more months.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Follow-up probiotic
- Probiotic (Experimental): This arm will receive probiotic for 6 months then will keep receiving probiotic for 6 more months.
  Interventions: Dietary Supplement: Probiotic; Dietary Supplement: Follow-up probiotic

INTERVENTIONS:
Dietary Supplement: Placebo — Intervention with a daily dose of placebo for 6 months
  Arms: Placebo
Dietary Supplement: Probiotic — Intervention with a daily dose of probiotic for 6 months
  Arms: Probiotic
Dietary Supplement: Follow-up probiotic — Intervention with a daily dose of probiotic for 6 months

SUMMARY:
A whole new research area studying the function of intestinal microorganisms, also known as gut microbiota, has emerged during the last decade. As a result, dietary supplementation with specific bacteria (or probiotics) holds great promise as a therapeutic strategy for a wide range of diseases, from obesity to anxiety and depression, all of which are major characteristics of Prader-Willi syndrome (PWS).

The main objective of the current proposal is to determine the effects of Bifidobacterium animalis subsp. lactis (strain BPL1) supplementation in children and young adults with PWS. Specifically, participants will receive placebo or BPL1 for 6 months, and then this phase will be followed by a 6-month extension period in which all participants will receive BPL1. This study will allow us to 1) determine the effects on fat mass and glucose metabolism; and 2) explore the effects on mental health symptoms by studying potential structural changes in the brain by magnetic resonance imaging (MRI) as well as using a number of psychiatric questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Prader-Willi Syndrome with genetic confirmation
* On a stable diet and medication regimen for at least the last two months before enrollment

Exclusion Criteria:

* Current enrollment in or discontinuation within the last 30 days from a clinical trial
* Patients with bariatric surgery in the last two years
* Patients with Type 2 Diabetes on insulin therapy
* Presence of other medical problems that would preclude study participation
* Unsuitable for inclusion in the study in the opinion of the investigator

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in percent body fat content | 6 months
  Body fat content will be measured by dual energy x-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Change in BMI and BMI z-score | Baseline, 6, and 12 months
  Weight and height will be combined to calculate changes in BMI and BMI z scores from all subjects will be assessed
Change in height (cm) | Baseline, 6, and 12 months
  Changes in height from subjects that have not yet reached final height will be measured.
Change in insulin sensitivity | Baseline, 6, and 12 months
  Fasting blood glucose and insulin concentrations will be combined to calculate HOMA-IR (Homeostatic Model Assessment for Insulin Resistance).
Change in lipid profile (triglyceride, cholesterol) | Baseline, 6, and 12 months
  Blood test after overnight fasting
Change in hyperphagia | Baseline, 6, and 12 months
  Measured by the validated Hyperphagia Questionnaire for Clinical Trials (HQ-CT), specific for subjects with Prader-Willi syndrome (scale 0-36, higher values indicate higher degree of hiperphagia). Parental or caregiver reported.
Change in Aberrant Behavior Checklist (ABC) score | Baseline, 6, and 12 months
  The Aberrant Behavior Checklist (ABC) is a 58-item questionnaire. It consists of five subscales: hyperactivity (0-48), lethargy (0-48), stereotypical behavior (0-21), irritability (0-45), and inappropriate speech (0-12). Higher scores indicate worse outcome. Parental or caregiver reported.
Change in Repetitive Behavior Scale (RBS) score | Baseline, 6, and 12 months
  The Repetitive Behavior Scale (RBS) measures repetitive behaviors that are related to autism. It consists of 43-items grouped in two different scores: higher-order (ritualistic, sameness, compulsive and restricted subscales; score 0-87) and lower-order (stereotypy and self-injury; score 0-42) repetitive behaviors. Higher scores indicate worse outcome. Parental or caregiver reported.
Change in Social Responsiveness Scale (SRS) score | Baseline, 6, and 12 months
  Measured by the validated Social Responsiveness Scale (SRS-2) which assesses autism-related symptoms focusing on social function. Higher values indicate worse outcome. A total score of 76 or higher is considered severe; a score between 66 and 75 is considered moderate; a score between 60 and 65 is considered mild; a score of 59 or lower is considered within normal limits. Parental or caregiver reported.
Change in Clinical Global Impression (GCI score) score | Baseline, 6, and 12 months
  Measured by the validated Clinical Global Impression Scale (CGI, scale 0-14, higher values indicate worse outcome). This toll will be completed by the clinician.

OTHER OUTCOMES:
Change in intestinal microbiota composition | Baseline, 6, and 12 months
  DNA isolated from fecal samples will be analyzed by sequencing the hypervariable region of the bacterial 16S gene.
Change in plasma metabolome | Baseline, 6, and 12 months
  Liquid chromatography coupled to mass spectrometry will be used to obtain a comprehensive metabolic profile of plasma samples
Changes in brain structural anatomy | Baseline, 6, and 12 months
  Subjects older that 12 years of age will undergo brain magnetic resonance imaging (MRI). Changes in orbitofrontal cortex, amygdala, hypothalamus, and total gray matter volume will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Ramon-Krauel, Principal Investigator — Hospital Sant Joan de Deu; Carles Lerin, PhD, Principal Investigator — Fundació Sant Joan de Déu
Locations (1):
- Hospital Sant Joan de Deu, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No